CLINICAL TRIAL: NCT03875001
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1358894 in Healthy Japanese Male Subjects (Double-blind, Randomised, Placebo-controlled Parallel Dose Group Design)
Brief Title: A Study About How Different Doses of BI 1358894 Are Taken up in the Body and How Well They Are Tolerated in Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1402-0008
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Experimental): For each dose group a placebo group was given matching placebo tablets, participants were randomized within each dose group in a 3:1 ratio (active drug:placebo), tablets taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Interventions: Drug: Placebo
- Dose group 1 - 50 mg BI 1358894 (Experimental): 2 film-coated tablets of 25 milligram (mg) BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Interventions: Drug: Dose group 1 - 50 mg BI 1358894
- Dose group 2 - 100 mg BI 1358894 (Experimental): 1 film-coated tablet of 100 milligram BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Interventions: Drug: Dose group 2 - 100 mg BI 1358894
- Dose group 3 - 200 mg BI 1358894 (Experimental): 2 film-coated tablets of 100 milligram BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Interventions: Drug: Dose group 3 - 200 mg BI 1358894

INTERVENTIONS:
Drug: Placebo — For each dose group a placebo group was given matching placebo tablets, participants were randomized within each dose group in a 3:1 ratio (active drug:placebo), tablets taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Arms: Placebo
Drug: Dose group 1 - 50 mg BI 1358894 — 2 film-coated tablets of 25 milligram (mg) BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Arms: Dose group 1 - 50 mg BI 1358894
Drug: Dose group 2 - 100 mg BI 1358894 — 1 film-coated tablet of 100 milligram BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Arms: Dose group 2 - 100 mg BI 1358894
Drug: Dose group 3 - 200 mg BI 1358894 — 2 film-coated tablets of 100 milligram BI 1358894 taken orally with ~240 milliliter of water 30 minutes after a standard high-fat, high-calorie meal (after an overnight fast of 10 hours).
  Arms: Dose group 3 - 200 mg BI 1358894

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1358894 in healthy male subjects following oral administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria:

  -- born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years (inclusive) at screening
* Body mass index (BMI) of 18.5 to 25.0 kg/m2 (inclusive) at screening
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use with their female partner, adequate contraception throughout the study and until three months after the last administration of trial medication. Adequate methods are:

  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), hormonal contraception (e.g., implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g., diaphragm with spermicide) Unprotected sexual intercourse with a pregnant female partner is not allowed throughout the study and until three months after the last administration of trial medication.

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* C-Reactive Protein (CRP) > upper limit of normal (ULN), erythrocyte sedimentation rate (ESR) ≥ 15 millimeters/hour, liver and kidney parameter above ULN, other laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including viral hepatitis, human immunodeficiency virus (HIV) and/or syphilis. (Subject with positive Hepatitis B core antibody will not be allowed to participate in this trial)
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 400 mL within 12 weeks or 200 mL within 30 days or plasma donation within 2 weeks prior to administration or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yoon J, Sharma V, Harada A. Safety, Tolerability, and Pharmacokinetics of Oral BI 1358894 in Healthy Japanese Male Volunteers. Clin Drug Investig. 2024 May;44(5):319-328. doi: 10.1007/s40261-024-01357-z. Epub 2024 Apr 24. PMID 38656736
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study tests the safety, tolerability and pharmacokinetics of single rising oral doses of BI 1358894 in healthy Japanese male subjects (double blind, randomised, placebo-controlled parallel dose group design)
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: This set included data from all subjects who received at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.1) | 26.3 (8.4) | 32.3 (8.4) | 29.8 (7.0) | 30.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug Related Adverse Events (AEs).
Description: Percentage of subjects with drug related adverse events (AEs).
Time Frame: Up to 14 days for 50 mg BI 1358894, 100 mg BI 1358894 and placebo. Up to 33 days for 200 mg BI 1358894.
Population: Treated set: This set included data from all subjects who received at least one dose of trial drug. The TS was used for safety analyses.
Measure: Number; unit: Percentage
Arm/Group | Placebo | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage | 0 | 0 | 16.7 | 33.3

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: AUC0-tz (area under the concentration-time curve of BI 1358894 in plasma over the time interval from the time of administration to the last quantifiable data time point tz).
Time Frame: 2 hours before and 0.17, 0.33, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 34, 48, 72, 96, 120, 144, 168*, 192, 240#, 336#, 504#, 672# hours following treatment. *only dose groups 1 and 2, #only dose group 3.
Population: Pharmacokinetic Set (PKS): This set included all subjects from the treated set who provide at least one Pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK, or due to PK non-evaluability, even subjects contributing with only 1 PK parameter were included in PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)* hour (h) / liter (L)
Arm/Group | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
Number analyzed (Participants) | 6 | 6 | 6
nanomole (nmol)* hour (h) / liter (L) | 6320 (15.0) | 13700 (23.5) | 32200 (26.0)

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)* hour (h) / liter (L)
Arm/Group | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
Number analyzed (Participants) | 6 | 6 | 6
nanomole (nmol)* hour (h) / liter (L) | 6960 (16.5) | 15800 (20.8) | 33600 (26.1)

4. Secondary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1358894 in plasma.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) / liter (L)
Arm/Group | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
Number analyzed (Participants) | 6 | 6 | 6
nanomole (nmol) / liter (L) | 224 (14.2) | 470 (22.3) | 904 (10.9)

ADVERSE EVENTS:
Time Frame: Up to 14 days for dose group 1, 2 (respectively 50 mg and 100 mg BI 1358894) and placebo and up to 33 days for dose group (200 mg BI 1358894).
Description: Treated set: This set included data from all subjects who received at least one dose of trial drug. The TS was used for safety analyses.
Arm/Group | Placebo | Dose Group 1 - 50 mg BI 1358894 | Dose Group 2 - 100 mg BI 1358894 | Dose Group 3 - 200 mg BI 1358894
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Dose Group 1 - 50 mg BI 1358894 (N=6) | Dose Group 2 - 100 mg BI 1358894 (N=6) | Dose Group 3 - 200 mg BI 1358894 (N=6)
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03875001/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03875001/SAP_001.pdf